CLINICAL TRIAL: NCT04481503
Title: Transthoracic Echocardiography of Cardiac Function of Parturients in Labor
Brief Title: Transthoracic Echocardiography of Ventricular Function of Parturients in Labor
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Leigh C. Hickerson, Assistant Professor of Anesthesiology, Dartmouth-Hitchcock Medical Center
Other Study IDs: D20144
Record Dates: First submitted 2020-07-14; First posted 2020-07-22 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Obstetric Labor Complications; Cardiovascular Diseases in Pregnancy; Cardiovascular Risk Factor
MeSH Terms: conditions — Obstetric Labor Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This echocardiography study will characterize heart structure and function during labor. Imaging of the heart during the stress of labor could increase detection of subclinical cardiovascular disease using advanced imaging techniques. Cardiac serum biomarkers and complication rates will also be measured and compared between patients with and without evidence of cardiovascular disease on echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* All healthy parturients 18 years of age or older with estimated gestation greater than or equal to 37 weeks who are expected to deliver during their hospitalization.
* During the echocardiographic exam, the patient must be in active labor with cervical dilation between 6-10 cm and contractions that are spaced less than 5 minutes apart.

Exclusion Criteria:

* Known functional or structural heart disease
* Previously diagnosed pulmonary hypertension.
* Comorbid disease other than diet controlled gestational diabetes, uncomplicated obesity, mild asthma and euthyroid patients with a history of hypo or hyperthyroidism.
* Parturients endorsing active use of non-prescription mind-altering drugs including cocaine, methamphetamine, or ketamine.
* Other non-inclusion criteria include inability to tolerate left lateral positioning either symptomatically or by fetal heart rate monitoring, suspected hypo-or hypercoagulable states that was not previously diagnosed, hemodynamic instability requiring >2 L crystalloid administration within 1 hour time frame after epidural placement or vasopressor administration of >15 mg ephedrine or >300 mcg phenylephrine administration within 1 hour after epidural placement.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Any pregnant patient, even if gender identity is male.
Study Population: Healthy women between 18 and 35 years of age with singleton pregnancy in active labor
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with an abnormal strain pattern as compared to parturients not in labor | During echocardiogram procedure
  Left ventricular strain
The proportion of patients with diastolic dysfunction as compared to parturients not in labor | During echocardiogram procedure
  Abnormal diastolic function

SECONDARY OUTCOMES:
Estimated right ventricular systolic pressure | During echocardiogram procedure
  Comparing estimated right ventricular systolic pressure between patients in active labor as compared to those who are not in active labor (mm Hg)

OTHER OUTCOMES:
Left ventricular systolic function | During echocardiogram procedure
  Simpson's method of discs motion abnormalities and diastolic function
Left ventricular myocardial performance index | During echocardiogram procedure
Total number of patients with the presence of regional wall motion abnormalities | During echocardiogram procedure
Total number of patients with abnormal global right ventricular dysfunction | During echocardiogram procedure
Right ventricular strain | During echocardiogram procedure
  %
Tricuspid annular plane systolic excursion | During echocardiogram procedure
  centimeters
Tissue doppler s' | During echocardiogram procedure
  cm/sec
Total number of maternal deaths within 0-42 days post-partum | 0 to 42 days post-partum
The number of patients with an identifiable Centers for Disease Control Severe Maternal Morbidity Identification complication post-partum | 0 to 42 days post-partum
  Acute myocardial infarction, aortic aneurysm, acute renal failure, adult respiratory distress syndrome, amniotic fluid embolism, cardiac arrest, ventricular fibrillation, conversion of cardiac rhythm, disseminated intravascular coagulation, eclampsia, heart failure, arrest during surgery or procedure, puerperal cerebrovascular disorders, pulmonary edema, aspiration, cardiopulmonary anesthesia complications, sepsis, shock, air or thrombotic embolism, blood product transfusion, hysterectomy, temporary tracheostomy, requiring ventilation
The number of patients with a pulse oximetry reading <90% after delivery | 0 to 42 days post-partum
The number of patients who required oxygen administration after delivery | 0 to 42 days post-partum
The number of patients who develop atrial fibrillation or premature atrial complexes | 0 to 42 days post-partum
The number of patients who develop a stroke | 0 to 42 days post-partum
  Stroke must be verified by imaging including either computed tomography or magnetic resonance imaging.
The number of patients with an elevation in transaminase levels during labor or after delivery | 0 to 42 days post-partum
Hospital length of stay | 0 to 42 days post-partum
  Total hours from admission to discharge
The number of patients requiring intensive care unit admission within 42 days post delivery | 0 to 42 days post-partum
Mortality within 42 days post delivery | 0 to 42 days post-partum
The number of patients with a post-partum diagnosis of post-partum hemorrhage | 0 to 42 days post-partum
The total number of patients who require additional uterotonic medications other than oxytocin after delivery | 0 to 42 days post-partum
  Medications include additional dosage of oxytocin above 3 units, methylergonovine, carboprost, tranexamic acid or misoprostol
The number of patients requiring a transfusion | 0 to 42 days post-partum
  Cell Saver, red blood cells, platelets, fresh frozen plasma, cryoprecipitate
Blood loss | 0 to 42 days post-partum
  Estimated and quantitated blood loss as well as the difference between pre-delivery hemoglobin and post-delivery lowest hemoglobin during admission
Number of patients requiring vasopressor after delivery to support blood pressure | 0 to 42 days post-partum
  phenylephrine, ephedrine, norepinephrine, epinephrine, vasopressin, inhaled nitrous oxide, inhaled epoprostenol
Activin A level | Less than 3 hours after echocardiogram procedure
Placental Growth Factor | Less than 3 hours after echocardiogram procedure
Soluble endoglin | Less than 3 hours after echocardiogram procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No